CLINICAL TRIAL: NCT05515042
Title: A Phase 2a Trial to Evaluate the Safety and Immunogenicity of COVID-19 Vaccine Strategies in HIV-infected and HIV-uninfected Adults.
Brief Title: Phase 2a Trial to Evaluate Safety and Immunogenicity of COVID-19 Vaccine Strategies in HIV-infected/Uninfected Adults.
Acronym: AUR1-8-341
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AUR1-8-341 CEPI; DOH-27-062022-4961 (Other: SANCTR)
Record Dates: First submitted 2022-07-11; First posted 2022-08-25 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: Vaccines
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1; Vaccines; BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, observer blind clinical trial. A total of 750 evaluable HIV-infected (660) and HIV-uninfected (90) adult participants meeting all entry criteria (all inclusion and no exclusion criteria) will be enrolled in 3 treatment strategies in 3 participant groups dependent on prior vaccination with a single dose Janssen (Group 1), 2 doses of Pfizer (Group 2) or no prior COVID-19 vaccination with evidence of prior SARS-CoV-2 infection (Group 3). A total of 300 participants per group will be enrolled in Groups 1 and 2 (255 HIV-infected and 45 HIV-uninfected per group), and 150 HIV-infected, unvaccinated participants in Group 3. Each treatment regimen (Vaccine Arm: A, B or C) will evaluate 250 participants. Groups 1 and 2 will enrol 85 HIV-infected and 15 HIV-uninfected per vaccine arm.
Who Masked: Participant, Investigator
Masking Description: Participants, investigators, and site staff (except for site pharmacists) will be blinded to participant treatment group assignment for the full duration of the study. Study product assignments are accessible to the site pharmacists and unblinded monitors who are required to know this information in order to ensure proper trial conduct. Any discussion of study product assignment between pharmacy staff and any other staff is prohibited. The DSMB members may be unblinded on request to treatment assignment, in order to conduct review of trial safety data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ad26.COV2.S (VAC31518, JNJ-78436735) Vaccine (Active Comparator): Description: The Ad26.COV2.Sis a recombinant, replication-defective adenovirus type 26 (Ad26) vector vaccine encoding the SARS-CoV-2 spike (S) glycoprotein.
  Dose: The Ad26.COV2.S drug product (DP) is supplied as a single-dose or multi-dose suspension (target DP titer is 1×1011 virus particles [vp]/mL or 2×1011 vp/mL) for intramuscular (IM) injection.
  Dosage Form: Sterile liquid suspension for injection Colourless to slightly yellow, clear to very opalescent suspension (pH 6-6.4).
  Packaging: The vaccine will be provided as a multi-dose vial with 5 doses per vial with a total volume of 2.5ml.
  Administration: Vaccination (5x10^10 vp dose) is given as a 0.5mL intramuscular injection into the deltoid muscle in the upper arm.
  Interventions: Drug: Ad26.COV2.S (VAC31518, JNJ-78436735) Vaccine, SARS-CoV-2 rS (CovovaxTM), BNT162b2 (Pfizer)
- SARS-CoV-2 rS (CovovaxTM) (Active Comparator): Description - SARS-CoV-2 rS (CovovaxTM): is a recombinant protein nanoparticle vaccine constructed from the SARS-CoV-2 full-length spike (S) glycoprotein co-formulated with Matrix-M1 adjuvant.
  Dose: Each 0.5ml of SARS-CoV-2 rS consists of 5μg of a recombinant nanoparticle spike protein plus 50 μg of Matrix-M1 adjuvant.
  Dosage Form: Suspension for injection COVOVAX™ is colourless to slightly yellow, clear to mildly opalescent, free to practically free from visible particles.
  Packaging: The vaccine will be supplied as a multi-dose vial containing 10 doses per vial Administration: Vaccinations are given as a 0.5mL intramuscular injection into the deltoid muscle in the upper arm
  Interventions: Drug: Ad26.COV2.S (VAC31518, JNJ-78436735) Vaccine, SARS-CoV-2 rS (CovovaxTM), BNT162b2 (Pfizer)
- BNT162b2 (Pfizer) (Comirnaty) (Active Comparator): Description: is a nucleoside-modified messenger RNA encoding the viral spike (S) glycoprotein of SARS-CoV-2. Vaccinations 30mcg (0.3mL) will be given as an intramuscular injection into the deltoid muscle in the upper arm.
  Dose: Each dose (0.3 mL) contains 30 micrograms of COVID-19 mRNA Vaccine. Dosage Form: White to off-white frozen suspension for Intramuscular (IM) injection Packaging: This vaccine will be supplied as a multidose vial and must be diluted with 0.9% Sodium Chloride USP before use. Each vial (0.45 mL) contains 6 doses of 0.3 mL after dilution.
  Administration: Comirnaty should be administered intramuscularly after dilution. Each dose must contain 0.3 mL of vaccine. The preferred site is the deltoid muscle of the upper arm
  Interventions: Drug: Ad26.COV2.S (VAC31518, JNJ-78436735) Vaccine, SARS-CoV-2 rS (CovovaxTM), BNT162b2 (Pfizer)

INTERVENTIONS:
Drug: Ad26.COV2.S (VAC31518, JNJ-78436735) Vaccine, SARS-CoV-2 rS (CovovaxTM), BNT162b2 (Pfizer) — As included in arm/group descriptions

SUMMARY:
This is a multicenter, randomized, observer blind clinical trial. A total of 750 evaluable HIV-infected (660) and HIV-uninfected (90) adult participants meeting all entry criteria (all inclusion and no exclusion criteria) will be enrolled in 3 treatment strategies in 3 participant groups dependent on prior vaccination with a single dose Janssen (Group 1), 2 doses of Pfizer (Group 2) or no prior COVID-19 vaccination with evidence of prior SARS-CoV-2 infection (Group 3) .A total of 300 participants per group will be enrolled in Groups 1 and 2 (255 HIV-infected and 45 HIV-uninfected per group), and 150 HIV-infected, unvaccinated participants in Group 3. Each treatment regimen (Vaccine Arm: A, B or C) will evaluate 250 participants. Groups 1 and 2 will enrol 85 HIV-infected and 15 HIV-uninfected per vaccine arm.

ELIGIBILITY:
Inclusion Criteria:

1. . Adult male or female aged 18 and above at the time of written informed consent
2. . Willing and able to give written informed consent
3. . HIV-infected persons on ART for at least three months prior to enrollment, or HIV-uninfected persons
4. . Able to provide evidence of completing a primary COVID-19 vaccination regimen with either a single dose of Ad26.COV2.S or two doses of BNT162b2 at least two months prior to enrolment, or HIV-infected with no prior COVID-19 vaccination and evidence of prior SAR-CoV-2 infection
5. . Residing in the vicinity of the clinical trial site and planning to remain in the area of the study for 12months
6. . Able and willing to participate for the duration of the study visits and follow-up
7. . Willing to provide verifiable identification (eg. Identity document, passport) at study entry and follow-up visits

Exclusion Criteria:

1. . Positive SARS-CoV-2 PCRor antigen detection test
2. . Persons with undocumented HIV status
3. . HIV-infected persons with CD4count <1 00 cells/mm3and/or Viral Load > 1000 copies/ml
4. . Known allergy or history of anaphylaxis or other serious adverse reactions to specific COVID-19 vaccine constituents
5. . History of capillary leak syndrome, thrombosis with thrombocytopenia syndrome (TTS), heparin-induced thrombocytopenia (HIT), history of any neurological disorders or seizures including Guillain-Barré syndrome, with the exception of febrile seizures during childhood
6. . Participants with acute illness (this does not include minor illnesses such as diarrhoea or mild upper respiratory tract infection) or body temperature ≥38.0ºC on Day 1 will be excluded from randomization at that time but may be rescheduled for randomization and/or vaccination at a later date.
7. . Participants who cannot communicate reliably with the investigator
8. . Pregnant or breastfeeding
9. . Women of childbearing potential who are not on an effective long-acting contraceptive method for at least 21 days prior to enrollment (date of signed informed consent) and not intending to continue contraception for up to 9 months post first vaccination.(See Section 10.5.1 below)
10. . Prior administration of an investigational coronavirus vaccine (for example, SARS-CoV-2, SARS-CoV, Middle East Respiratory Syndrome [MERS-CoV] vaccine), except for participants of the Sisonke trial
11. . Prior administration of any SARS-CoV-2 vaccine boost
12. . Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment
13. . History of harmful substance or alcohol use within the past 2 years. This exclusion does not apply to cannabis use.
14. . Receipt of:

    1. . Systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to the day of randomization (for corticosteroids, ≥20 mg/day prednisone equivalent). Topical tacrolimus is allowed if not used within 14 days prior to the day of randomization. Inhaled, nasal, and topical steroids are allowed.
    2. . Intravenous blood products (red cells, platelets, immunoglobulins, monoclonal antibodies specific for SARS-CoV-2) within 3 months prior to enrollment
    3. . Experimental vaccine within the past 6 months before first vaccination
    4. . Any inactivated vaccines received within 14 days prior to first vaccination or planned within 14 days of first vaccination, or live attenuated vaccines received with 30 days prior to the first vaccination or planned within 30 days of the first vaccination.
15. . Participated in an interventional clinical study within 28 days prior to the Screening Visit (Day 1) or plans to do so while participating in this study.
16. . Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective and Endpoint/Outcome 1: | 14 Months
  In HIV-infected persons, to determine whether each boost vaccine regimen adequately boosts humoral immune responses (D15), overall and by prior vaccine regimen. In this case humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 1:
  • Geometric mean value of SARS CoV-2 spike RBD protein-specific binding antibody (bAb) at baseline and D15, where bAb is measured from serum using an ELISA-based antibody binding assay to the SARS-CoV-2 RBD protein. The ELISA-based antibody binding assay to the SARS-CoV-2 RBD protein will be used to measure the serum bAb concentrations. The bAb concentrations will be derived from the half-maximal Effective Concentration (EC50) and the Area under the curve (AUC), and summarised as the Geometric mean value of bAb
Primary Objective and Endpoint/Outcome 2: | 14 Months
  In HIV-infected persons, to determine whether each boost vaccine regimen adequately boosts humoral immune responses (D15), overall and by prior vaccine regimen. In this case humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 2:
  • Geometric mean value of SARS CoV-2-specific neutralizing antibody (nAb) at baseline and D15 where nAb is measured from serum using a pseudovirus neutralizing assay. The SARS-CoV-2 VSV pseudotyped virus-based assay will be used measure the serum nAb concentrations. The nAb concentrations will be derived from Half-maximal inhibitory concentration (IC50), and summarised as the Geometric mean value of nAb

SECONDARY OUTCOMES:
Secondary Objective 1 and Endpoint/Outcome 1: | 14 Months
  In HIV-infected persons, to compare between Vaccine Arms (A, B, or C) humoral immune responses post boost vaccination (Day 15 and Months 6 and 12), overall and stratified by primary vaccination regimen, duration since primary vaccination, and age group. In this case humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 1:
  • The ELISA-based antibody binding assay to the SARS-CoV-2 RBD protein will be used to measure the serum bAb concentrations. Geometric mean value of SARS CoV-2 spike RBD protein-specific binding antibody (bAb) at Day 15 and Months 6 and 12 is determined from the half-maximal Effective Concentration (EC50) and the Area under the curve (AUC)
Secondary Objective 1 and Endpoint/Outcome 2: | 14 Months
  In HIV-infected persons, to compare between Vaccine Arms (A, B, or C) humoral immune responses post boost vaccination (Day 15 and Months 6 and 12), overall and stratified by primary vaccination regimen, duration since primary vaccination, and age group. In this case humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 2:
  • The SARS-CoV-2 VSV pseudotyped virus-based assay will be used measure the serum nAb concentrations. Geometric mean value of SARS CoV-2-specific neutralizing antibody (nAb) at Day 15 and Months 6 and 12 as measured by the half-maximal inhibitory concentration (IC50)
Secondary Objective 2 and Endpoint/Outcome 1: | 14 Months
  In HIV-infected persons, to describe the safety of each COVID-19 boost vaccine regimen. In this study safety is measured by moderate or severe solicited local and systemic adverse event (AE), serious adverse events (SAEs), medically attended AEs (MAAEs), or adverse events of special interest (AESI)
  Endpoint/Outcome 1:
  • Solicited local and systemic adverse events (AEs) within 7 days after each vaccine dose. The proportion of participants with at least one moderate or severe solicited local and systemic adverse event (AE) within 7 days after each vaccine dose, presented by study arm
Secondary Objective 2 and Endpoint/Outcome 2: | 14 Months
  In HIV-infected persons, to describe the safety of each COVID-19 boost vaccine regimen. In this study safety is measured by moderate or severe solicited local and systemic adverse event (AE), serious adverse events (SAEs), medically attended AEs (MAAEs), or adverse events of special interest (AESI)
  Endpoint/Outcome 2:
  • Unsolicited AEs within 28 days after each vaccine dose. The proportion of participants with at least one unsolicited AE within 28 days after each vaccine dose presented by study arm and stratified per study group
Secondary Objective 2 and Endpoint/Outcome 3: | 14 Months
  In HIV-infected persons, to describe the safety of each COVID-19 boost vaccine regimen. In this study safety is measured by moderate or severe solicited local and systemic adverse event (AE), serious adverse events (SAEs), medically attended AEs (MAAEs), or adverse events of special interest (AESI)
  Endpoint/Outcome 3:
  • The frequency of Serious adverse events (SAEs), medically attended AEs (MAAEs), or adverse events of special interest (AESI) from the first vaccine dose for up to 12 months after the last vaccine dose, presented by study arm and stratified per study group
Secondary Objective 3 and Endpoint/Outcome 1: | 14 Months
  In HIV-infected persons, to compare between Vaccine Arms (A, B, or C) the cellular immunogenicity post boost (D15 and months six and twelve), overall and stratified by primary vaccination regimen, duration since primary vaccination and age group. In this study cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
  Endpoint/Outcome 1:
  • The SARS CoV-2 specific T-cell responses will be measured by the IFN-gamma ELISpot assay. In this study the outcome measure for IFN-gamma ELISpot is Spot Forming Units per 10^6 cells.
Secondary Objective 3 and Endpoint/Outcome 2: | 14 Months
  In HIV-infected persons, to compare between Vaccine Arms (A, B, or C) the cellular immunogenicity post boost (D15 and months six and twelve), overall and stratified by primary vaccination regimen, duration since primary vaccination and age group. In this study cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
  Endpoint/Outcome 2:
  • The SARS CoV-2 specific CD4+ and CD8+ T-cell response will be measured by flow cytometry. The outcome measure for flow cytometry is the percentage T cell responses for the following cytokines: IFN-γ, IL-2, TNF-α and Granzyme B

OTHER OUTCOMES:
Exploratory Objective 1 and Endpoint/Outcome 1: | 14 Months
  To examine the immunologic imprint and pre-existing cross-reactive T-cell memory on vaccine induced antibody and T-cell responses in HIV-infected and HIV-uninfected participants. The coronavirus antigen microarray (CoVAM), Human virome-wide peptide library (PepSeq) and the Activation-induced T-cell marker assay (AIM) assay will be used to measure the immunologic imprint and pre-existing of cross-reactive T-cell memory on vaccine induced antibody and T-cell responses.
  Endpoint/Outcome 1:
  • Influence of pre-existing immunity on vaccine induced antibody and T-cell responses using coronavirus antigen microarray (CoVAM). The CoVAM outcome measure is the composite SARS-CoV-2 IgG mean fluorescence intensity (MFI) +/-95% CI
Exploratory Objective 1 and Endpoint/Outcome 2: | 14 Months
  To examine the immunologic imprint and pre-existing cross-reactive T-cell memory on vaccine induced antibody and T-cell responses in HIV-infected and HIV-uninfected participants. The coronavirus antigen microarray (CoVAM), Human virome-wide peptide library (PepSeq) and the Activation-induced T-cell marker assay (AIM) assay will be used to measure the immunologic imprint and pre-existing of cross-reactive T-cell memory on vaccine induced antibody and T-cell responses.
  Endpoint/Outcome 2:
  • Influence of pre-existing immunity on vaccine induced antibody and T-cell responses using coronavirus antigen microarray PepSeq assay. The PepSeq outcome measure ins the descriptive analysis of the frequency, kinetics and type of conserved, non-conserved and cross-reactive spike-specific epitopes
Exploratory Objective 1 and Endpoint/Outcome 3: | 14 Months
  To examine the immunologic imprint and pre-existing cross-reactive T-cell memory on vaccine induced antibody and T-cell responses in HIV-infected and HIV-uninfected participants. The coronavirus antigen microarray (CoVAM), Human virome-wide peptide library (PepSeq) and the Activation-induced T-cell marker assay (AIM) assay will be used to measure the immunologic imprint and pre-existing of cross-reactive T-cell memory on vaccine induced antibody and T-cell responses.
  Endpoint/Outcome 3:
  • The activation status of CD4+ and CD8+ T-cells using the AIM assay at baseline. The AIM assay outcome measure is the Geometric mean +/- 95% CI of AIM+ (OX40+CD137+) CD4+ and (CD69+CD137+) CD8+ T cells
Exploratory Objective 2 and Endpoint/Outcome 1: | 14 Months
  To describe COVID-19 infection and disease in trial participants.
  Endpoint/Outcome 1:
  • Number of participants with SARS CoV-2 infection (nucleocapsid antibody positive) will be determined using the SARS-CoV-2 Real Time (RT) PCR assay. The Thermofischer TaqPathTM COVID-19 CE-IVD RT-PCR will used to determine SARS CoV-2 infection. Participants with a positive RT PCR result will be regarded as SARS CoV-2 infected. The outcome measure of the RT PCR assay is the cycle threshold (Ct) values.
Exploratory Objective 2 and Endpoint/Outcome 2: | 14 Months
  To describe COVID-19 infection and disease in trial participants.
  Endpoint/Outcome 2:
  • Number of participants with COVID-19 disease (RT PCR positive) will be determined using the nucleocapsid-specific binding antibody. In this case the Abbott SARS-CoV-2 IgG chemiluminescent assay will be used to measure the serum nucleocapsid antibody concentrations. Participants with a positive a nucleocapsid antibody result will be regarded as SARS CoV-2 infected. The outcome measure of the Abbott SARS-CoV-2 IgG chemiluminescent assay is the N SARS-CoV-2 N protein IgG Index S/C.
Exploratory Objective 3 and Endpoint/Outcome: | 14 Months
  To characterize B-cell function and specificity in HIV-infected and HIV-uninfected participants post vaccination. In this case B-cell sorting and antibody sequencing will be used to determine the immunogenetic profiles of antibody lineages. Differences in the immunogenetic profiles of antibody lineages (including germline gene usage, percent somatic hypermutation and CDRH3 length), Clonal expansion and affinity maturation of memory B cells, Convergence of SARS-CoV-2 directed "public" antibody repertoires shared by participants.
  Endpoint/Outcome:
  The outcome will be B-cell germline gene usage, percent (%) somatic hypermutation and CDRH3 length
Exploratory Objective 4 and Endpoint/Outcome 1: | 14 Months
  To compare humoral and cellular immune responses post boost vaccination (Day 15 and months 6 and 12) among participants with or without prior SARS-CoV-2 infection in HIV-infected and HIV-uninfected participants, overall and by Vaccine Arm. Humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 1:
  • Geometric mean value of SARS CoV-2 spike RBD protein-specific binding antibody (bAb) at baseline and D15, month 6 and month 12 where bAb is measured from serum using an ELISA-based antibody binding assay to the SARS-CoV-2 RBD protein. Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells
Exploratory Objective 4 and Endpoint/Outcome 2: | 14 Months
  To compare humoral and cellular immune responses post boost vaccination (Day 15 and months 6 and 12) among participants with or without prior SARS-CoV-2 infection in HIV-infected and HIV-uninfected participants, overall and by Vaccine Arm. Humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 2:
  • Geometric mean value of SARS CoV-2-specific neutralizing antibody (nAb) at baseline, D15, month 6 and month 12 where nAb is measured from serum using a pseudovirus neutralizing assay. Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells
Exploratory Objective 4 and Endpoint/Outcome 3: | 14 Months
  To compare humoral and cellular immune responses post boost vaccination (Day 15 and months 6 and 12) among participants with or without prior SARS-CoV-2 infection in HIV-infected and HIV-uninfected participants, overall and by Vaccine Arm. Humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb).
  Endpoint/Outcome 3:
  • Mean SARS CoV-2 specific CD4+ and CD8+ T-cell responses by intracellular cytokine staining at Day 15 and months 6 and 12.
Exploratory Objective 5 and Endpoint/Outcome 1: | 14 Months
  To describe among HIV-infected, unvaccinated, participants with prior SARS-C0V-2 infection, humoral and cellular immune responses post boost vaccination (Day 15 and months 6 and 12), overall and by Vaccine Arm. Humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb). Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
  Endpoint/Outcome 1:
  • Geometric mean value of SARS CoV-2 spike RBD protein-specific binding antibody (bAb) at baseline and D15, month 6 and month 12 where bAb is measured from serum using an ELISA-based antibody binding assay to the SARS-CoV-2 RBD protein. Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
Exploratory Objective 5 and Endpoint/Outcome 2: | 14 Months
  To describe among HIV-infected, unvaccinated, participants with prior SARS-C0V-2 infection, humoral and cellular immune responses post boost vaccination (Day 15 and months 6 and 12), overall and by Vaccine Arm. Humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb). Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
  Endpoint/Outcome 2:
  • Geometric mean value of SARS CoV-2-specific neutralizing antibody (nAb) at baseline, D15, month 6 and month 12 where nAb is measured from serum using a pseudovirus neutralizing assay. Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
Exploratory Objective 5 and Endpoint/Outcome 3: | 14 Months
  To describe among HIV-infected, unvaccinated, participants with prior SARS-C0V-2 infection, humoral and cellular immune responses post boost vaccination (Day 15 and months 6 and 12), overall and by Vaccine Arm. Humoral response refers to SARS CoV-2 spike RBD protein-specific binding antibody (bAb) IgG and SARS CoV-2-specific neutralizing antibody (nAb). Cellular immunogenicity is measured by SARS CoV-2 specific CD4+ and CD8+ T-cell responses using ELISpot and flow cytometry from peripheral blood mononuclear cells.
  Endpoint/Outcome 3:
  • Mean SARS CoV-2 specific CD4+ and CD8+ T-cell responses by intracellular cytokine staining at Day 15 and months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Prof Gavin Churchyard, PhD, Principal Investigator — The Aurum Institute NPC
Locations (5):
- South Africa (5):
  - The Aurum Institute: Pretoria Clinical Research Centre, Pretoria, Gauteng
  - The Aurum Institute: Tembisa Clinical Research Centre, Clinic 4, Tembisa, Gauteng
  - The Aurum Institute: Tembisa Clinical Research Centre, Tembisa, Gauteng
  - The Aurum Institute: Gavin J Churchyard Legacy Centre, Klerksdorp, North West
  - The Aurum Institute: Rustenburg Clinical Research Centre, Rustenburg, North West

IPD SHARING:
Plan to Share IPD: Yes
The applicants are committed to the open science practice and will ensure rapid sharing of research results with scientific communities, policy makers and public of interest through peer-reviewed journal, national and international conferences. All publications will adopt open access principles based on the gold and green models. The study team will prepare a dissemination plan for study updates and results dissemination to high level stakeholders (IECs, Ministries of Health, NDR, government officials and international stakeholders). Study updates will be communicated to participants, CAB, study staff and other key stakeholders (trial networks, health advocates) timeously. The proposed trial will be registered at the Clinicaltrials.gov and South African Clinical Trials Register (SANCTR). Investigators will write and review the interim analysis and final analysis reports and publications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Quarter 4 2023
Access Criteria: Publication in Open Access Repositories will ensure that publications are publicly discoverable, accessible, and re-usable as soon as possible. After appropriate data clearance, and where appropriate IP arrangements have been made, we will make use of pre-print archives such as bioRxiv/medRxiv or Zenodo to stimulate immediate exchange and discussion of results, prior to peer-reviewed publication. Any further manuscripts, abstracts, press releases and publications that may arise from the study will be reviewed by all investigators. A full publication plan will be developed with all investigators and the funder once the study results are available.